CLINICAL TRIAL: NCT06977568
Title: A Phase 2, Randomized, Open-Label, Two-Arm Study to Evaluate a Procedure for Intra-Articular Injection of ZILRETTA Versus Triamcinolone Acetonide, Immediate Release (TCA-IR) in Subjects With Osteoarthritis of the Hip
Brief Title: A Study to Evaluate an Intra-Articular Injection of ZILRETTA Versus Triamcinolone Acetonide, Immediate Release in Subjects With Osteoarthritis of the Hip
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped due to business decision and lack of enrollment. There were no safety concerns.
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 006-C-202
Record Dates: First submitted 2025-05-07; First posted 2025-05-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis of Hip
Keywords: ZILRETTA; Osteoarthritis of Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to 1 of the 2 treatment arms: 1:1 across the 2 study drugs (ZILRETTA and TCA-IR) and a 1:1 ratio within each needle-gauge size (20- and 22-G) (approximately 8 subjects assigned to Arm 1A, approximately 8 subjects assigned to Arm 1B, approximately 8 subjects assigned to Arm 2A, and approximately 8 subjects assigned to Arm 2B)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1A: ZILRETTA and 20G Needle (Experimental): 32mg ZILRETTA and 20-G Spinal Needle
  Interventions: Drug: Zilretta
- 1B ZILRETTA and 22G Needle (Experimental): 32mg ZILRETTA and 22-G Spinal Needle
  Interventions: Drug: Zilretta
- 2A TCA-IR and 20G Needle (Active Comparator): 40mg TCA-IR and 20G Spinal Needle
  Interventions: Drug: Triamcinolone Acetonide
- 2B TCA-IR and 22G Needle (Active Comparator): 40mg TCA-IR and 22G Needle
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Zilretta — triamcinolone acetonide, extended release injectable suspension
  Other Names: triamcinolone acetonide, extended release injectable suspension
  Arms: 1A: ZILRETTA and 20G Needle; 1B ZILRETTA and 22G Needle
Drug: Triamcinolone Acetonide — Triamcinolone Acetonide, Immediate Release (TCA-IR)
  Other Names: Triamcinolone Acetonide, Immediate Release; TCA-IR
  Arms: 2A TCA-IR and 20G Needle; 2B TCA-IR and 22G Needle

SUMMARY:
The goal of this clinical trial is to evaluate an injection procedure for the investigational drug in people with Osteoarthritis of the Hip. The Sponsor is conducting this research to evaluate successful injections in the hip by using two different needle sizes.

ELIGIBILITY:
Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Participants must provide written informed consent prior to initiating any study specific procedures.
2. Participants must be willing and able to comply with the study procedures and visit schedule and to follow verbal and written instructions.
3. Participants must be male or female and 50 to 80 years old, inclusive, on the day of consent.
4. Participants must have a body mass index (BMI) ≤40 kg/m2 at Screening.
5. Participants must exhibit symptoms associated with unilateral or bilateral hip OA for at least 6 months prior to Screening.
6. Participants with unilateral or bilateral hip pain must have a 24-hour average pain score (based on a numerical rating scale [NRS]) between ≥5.0 and ≤9.0 for the index hip and <5 in contralateral hip at Screening.
7. Participants must have K-L Grade 1, 2, 3, or 4 in the index hip (ie, the hip identified by the Investigator as appropriate for injection) confirmed by X-ray obtained during Screening or within ≤6 months prior to the Screening visit.
8. Participants must have an index hip examination indicating the index hip and the intended injection site area must be free of any signs of local or joint infection at Day 1/Baseline. Participants must also not have a history of infection (eg, osteomyelitis) in the index hip or injection site.
9. Sexually active participants of child-bearing potential (POCBP; defined as neither surgically sterile nor postmenopausal, ie, age >45 years and no menstrual periods for at least 1 year without an alternative medical cause) must agree to use, from Screening through 14 weeks postinjection for biologically female participants and through 23 weeks postinjection for biologically male participants, a highly effective method of contraception, defined as one of the following: abstinence; oral, injected, or implanted hormonal methods of contraception; intrauterine device or intrauterine contraceptive system; condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; or sexual intercourse only with biological male ≥6 months post-vasectomy.

5.4. Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

1. Participants who are pregnant, nursing, lactating, or plan to become, or their partner plans to become, pregnant during the study.
2. Participants with a history of hypersensitivity to triamcinolone acetonide, PLGA, or lidocaine.
3. Participants with hypersensitivity or allergy to Omnipaque 300 or iodine.
4. Participants with a contraindication to the use of acetaminophen/paracetamol (allowed rescue pain medicine) per National Product Labeling and Investigator's judgment.
5. Participants currently taking coumadin or have taken coumadin for ≥3 weeks prior to Day 1/Baseline.
6. Participants with a history of or active significant concomitant illness (known or suspected) including, but not limited to:

   * Inflammatory joint disease, eg, rheumatoid arthritis, seronegative spondyloarthropathy, ankylosing spondylitis, psoriatic arthritis, reactive arthritis, inflammatory-bowel disease-associated inflammatory arthritis.
   * Systemic inflammatory disease, eg, polymyalgia rheumatica, systemic lupus erythematosus.
   * Sarcoidosis or amyloidosis.
   * Cushing's syndrome.
   * Malignancy requiring systemic therapy within the past 5 years (excludes basal cell carcinoma or cervical cancer treated only with surgical removal more than 1 year prior).
   * Other autoimmune disease.
7. Participants who have had any previous substantial hip injury (eg, hip dislocation, partial or complete hip fraction), which resulted in functional limitation or immobilization within 3 months prior to Screening.
8. Participants who have had prior surgery of the index hip either open or arthroscopic within 6 months of Screening.
9. Participants with any retained hardware or foreign body in the index hip.
10. Participants with an index hip with major dysplasia or congenital abnormality, osteochondritis dissecans, acromegaly, ochronosis, hemochromatosis, Wilson's disease, primary osteochondromatosis, chondrolysis from a pain pump, or a history of avascular necrosis with secondary OA.
11. Participants with a diagnosis of other disorders in the index hip that can cause pain or any concurrent chronic joint, muscle, or nerve pain condition within 1 month prior to Screening (participant self-report acceptable), including but not limited to, back spine pain or conditions causing femoral nerve, obturator nerve, and sciatic nerve injury/entrapment; trochanteric bursitis; diabetic neuropathy of lower extremities; post-herpetic neuralgia; post-stroke pain; or fibromyalgia that may affect sensation of the index hip.
12. Participants who have used corticosteroid injections in the index hip (IA, intrabursal, or intratendinous) or intravenous (IV), intramuscular (IM), or oral within 3 months of Screening. Also, participants who will require any systemic steroid use (oral, IV, or IM) while they are in the study are ineligible. Steroid injections in any other joint outside the index hip joint during the study are permitted.
13. Participants who have received IA treatment in the index hip with any of the following agents within the 6 months or 5 half-lives prior to Screening: any biologic agent (eg, platelet-rich plasma, stem cells, prolotherapy, amniotic fluid) or hyaluronic acid (within 3 months prior to Screening) (investigational or marketed).
14. Participants with a history of or evidence of active or latent systemic fungal or mycobacterial infection (including tuberculosis), or of ocular herpes simplex.
15. Participants who have received a live vaccine (eg, measles, mumps, and rubella [MMR], varicella, influenza [nasal spray version only], Bacillus Calmette-Guérin [BCG], and polio) within 3 months prior to Screening.
16. Participants who have received an inactivated vaccination (eg, flu, COVID, tetanus, tetanus/diphtheria/pertussis [Tdap], hepatitis A) within 1 week prior to Screening and local injection pain has not resolved.
17. Participants with diabetes mellitus with hemoglobin A1c (HbA1c) >8.5% at Screening.
18. Participants with evidence of positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Hepatitis B virus (HBV) immune participants (ie, HBsAg-negative and hepatitis B antibody-positive) may, however, be included.

    Note: Participants who are negative for HBsAg, but positive for HBcAb, would be considered eligible if the absence of HBV DNA is confirmed by HBV DNA polymerase chain reaction reflex testing.
19. Participants with chronic hepatitis C virus (HCV) (ie, positive HCV antibody [HCVAb] and HCV RNA).

    Note: Participants who are HCVAb-positive without evidence of HCV RNA may be considered eligible (spontaneous viral clearance or previously treated and cured [defined as no evidence of HCV RNA at least 3 months prior to Day 1/Baseline]).
20. Participants with laboratory evidence of infection with human immunodeficiency virus (HIV).
21. Participants who have any infection requiring parenteral antibiotics within 4 weeks of Day 1/Baseline or oral antibiotics within 2 weeks of Day 1/Baseline.
22. Participants with active substance use disorder (drugs or alcohol) or history of substance use disorder within 12 months prior to Screening. Positive amphetamine results due to prescribed attention deficit/hyperactivity disorder (ADHD) medications with at least 6 months of stable dosing is permitted.
23. Participants who use muscle relaxants (eg, cyclobenzaprine, tetrazepam, and diazepam) or oral/topical therapies (eg, nonsteroidal anti-inflammatory drugs [NSAIDs], cannabidiol [CBD] oil, capsaicin, lidocaine patches, or other local treatments) applied to the index hip within 1 month prior to Screening or within 5 half-lives of last dose.
24. Participants who use selective serotonin reuptake inhibitors (SSRIs)/serotonin and norepinephrine reuptake inhibitors (SNRIs) (eg, fluoxetine, fluvoxamine, citalopram, escitalopram, sertraline, duloxetine, venlafaxine, and milnacipran) if the dose is not stable for at least 3 months prior to Screening. Participant must remain on a stable dose throughout the study.
25. Participants using immunomodulators, immunosuppressives, or chemotherapeutic agents or have used any within 5 years of Screening.
26. Participants using any other investigational drug, biologic, or device or have used any within 3 months of Screening.
27. Participants who cannot washout prohibited medications (eg, opioids, other analgesics, and tetrahydrocannabinol [THC]- and CBD-containing products) or restricted medications.
28. Participants who have any abnormal laboratory value(s) at Screening that, in the opinion of the Investigator (or other authorized clinical staff), precludes study participation.
29. Participants with any other clinically significant acute or chronic pain condition that, in the judgment of the Investigator and in consultation with the MM and/or sponsor, would or could compromise (or convey increased risk of) participant safety, limit the participant's ability to complete the study, and/or compromise the objectives of the study.
30. Participants with any other clinically significant acute or chronic medical conditions (eg, autoimmune disorder; asthma/chronic obstructive pulmonary disease [COPD], or allergies requiring steroid use; bleeding disorder; other major hematological conditions, cardiac, renal, metabolic, gastrointestinal, neurologic, or psychiatric disease) that, in the judgment of the Investigator and/or in consultation with the MM, would preclude the use of the study drug or IA corticosteroids or that could compromise (or convey increased risk of) participant safety, limit the participant's ability to complete the study, and/or compromise the objectives of the study.
31. Participants are the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other staff, or relative thereof directly involved in the conduct of the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-07-25 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Assessment of Successful Hip injection Rate | Day 1
  The assessment of successful hip injection rate (injection of the full dose) for ZILRETTA and TCA-IR based on the 2 different needle-gauges

SECONDARY OUTCOMES:
TEAE, AESIs, SAEs | From Day 1 through Week 12
  Incidence of related treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), and serious adverse events (SAEs) from Day 1 through Week 12 for ZILRETTA and TCA-IR.
Change in 24-hour average pain score | Change from Baseline to Week 1, Week 4, Week 8, and Week 12
  Change from Baseline at Weeks 1, 4, 8, and 12 in the 24-hour average pain score (based on a numerical rating scale [NRS]) for ZILRETTA and TCA-IR . Average pain score is rated on a numerical scale between 0 (no pain) and 10 (worst possible pain).
Change in HOOS Survey | Change from Baseline to Week 1, Week 4, Week 8, and Week 12
  Change from Baseline at Weeks 1, 4, 8, and 12 on the Hip Disability and Osteoarthritis Outcome Score (HOOS) total score and all subscales for ZILRETTA and TCA-IR. The HOOS includes 40 questions with five possible responses, graded from 0 to 4. Total HOOS to be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Nino Joy, Study Director — Pacira Pharmaceuticals, Inc; Martin Ferrillo, Principal Investigator — Medical Pain Management Services, PLLC
Locations (1):
- Medical Pain Management Services PLLC, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Based on written request for IPD sharing.
Time Frame: Based on written request.
Access Criteria: Based on written request.